



## Evaluating The Effect of Probiotics on Oral Health Status and its Influence on The Gingival Disease and Halitosis in Iraq

Research ethics: patient consent form

Master Student: Baydaa Abdulqahar Younus

Date: 5 \January\2025

## **RESEARCH ETHICS: PATIENT CONSENT FORM**

**Study Number: MUPRV0013** 

Patient Identification Number for this trial: No. 1



Title of Project: Evaluating the Effect of Probiotics on Oral Health Status and its Influence on the Gingival Disease and Halitosis in Iraq

Principle investigator: Baydaa Abdulqahar Younus

- I confirm that I have read and understand the information sheet dated for the above study and have had the opportunity to ask questions.
- I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected.
- I understand that sections of any of my medical notes may be looked at by responsible individuals from regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records
- I agree to take part in the above study.

| Name of participant | Date | | Signature |
|-------------------------------|------|------|-----------|
| Name of Person taking consent | | Date | Signature |